CLINICAL TRIAL: NCT04236063
Title: Rehabilitation Needs of the Malaysian Haematological Cancer Survivors Through a Single Centre Experience
Brief Title: Rehabilitation Needs of the Malaysian Haematological Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chan Soo Chin, Senior Lecturer and Rehabilitation Physicians, University of Malaya
Other Study IDs: 201945-7310
Record Dates: First submitted 2019-09-23; First posted 2020-01-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Haematological Malignancy; Leukemia, Acute; Lymphoma; Myeloma Multiple; Blood Cancer; Quality of Life
Keywords: Cross sectional study
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haematological malignancy: Patients with haematological malignancy
  Interventions: Other: WHODAS 2.0 Questionnaire

INTERVENTIONS:
Other: WHODAS 2.0 Questionnaire — 36-item WHODAS 2.0 questionnaire will be used for each patient to identify difficulty faced by patient over past 30 days from the day of interview

SUMMARY:
Many cancers are being treated more effectively nowadays due to the raised awareness and early detection as well as advancement in researches and technology. Despite the rising number of cancer survivors in the coming years, these survivors are still plagued by the poor quality of life due to physical and psychological impairment. According to the National Cancer Registry Report from 2007-2011, haematological cancer is one of the ten most common cancers in Malaysian population. Many haematological cancer survivors in Malaysia are reportedly having poor quality of life due to multiple physical and emotional impairments which leads to further disability in life. It is thus an important effort to identify the rehabilitation needs in these cancer survivors to implement alternatives to improve the disease outcome through cancer rehabilitation.

DETAILED DESCRIPTION:
A cross-sectional questionnaire-based study will be employed to identify the rehabilitation needs and predictors of needs in outpatient hemato-oncological cohort at UMMC Hemato-oncology Clinic for 12 months. The validated questionnaire employed evaluates the potential disabilities that could affect the aforementioned patients in domains such as communication, independence in mobility, self-care, social participation, handling relationships and domestic activity of daily living a month prior to the survey.

Participants of age between 18 to 80 years old, diagnosed with haemato-oncological illnesses will be screened; excluding potential participants who are too ill or cannot understand English, Malay, or Chinese; to be recruited in the research.

Based on the findings from the analysis, rehabilitation needs could be tailored accordingly to improve quality of life of these patients

ELIGIBILITY:
Inclusion Criteria:

* patient with haematological malignancy
* agreeable to participate in the interview

Exclusion Criteria:

* ill at the time of follow up
* unable to understand English, Malay or Chinese
* refuse to be interviewed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with haematological malignancy under follow up at UMMC Haemato-oncology clinic
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 | 30 days ago from interview date
  WHODAS 2.0 is a practical, generic assessment tool that measures health and disability at population level or in clinical practice. It identifies possible disabilities in 6 domains of life namely Cognitive, Mobility, Self Care, Relationship, Life Activities and Participation. In view of its resemblance to the International Classification of Functioning, Disability and Health (ICF) model, direct identification of functioning and disability separately from the disease condition could be done.
  Each domain has few sets of questions pertaining to the activities; the responses and scores of each question are divided into none (0), mild (1), moderate (2), severe (3) and extremely cannot do (4). The scores from each domain will be summed and higher scores signifies higher disability status.

SECONDARY OUTCOMES:
Identifying patients who are at risk of disability from haemato-oncological illness | 30 days ago from interview date
  Disability outcomes of different groups of patients (of demographics and diagnosis) were analyzed using SPSS program and identification of patients who were vulnerable to haematological cancers were done using ANOVA test.

CONTACTS AND LOCATIONS:
Overall Officials: SOO CHIN CHAN, MASTERS, Principal Investigator — SENIOR LECTURER AND REHABILITATION PHYSICIAN; ANWAR SUHAIMI, MASTERS, Principal Investigator — SENIOR LECTURER AND REHABILITATION PHYSICIAN
Locations (1):
- University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Okamura H. Importance of rehabilitation in cancer treatment and palliative medicine. Jpn J Clin Oncol. 2011 Jun;41(6):733-8. doi: 10.1093/jjco/hyr061. PMID 21622762
- [Result] Allart-Vorelli P, Porro B, Baguet F, Michel A, Cousson-Gelie F. Haematological cancer and quality of life: a systematic literature review. Blood Cancer J. 2015 Apr 24;5(4):e305. doi: 10.1038/bcj.2015.29. PMID 25909835
- [Result] Priscilla D, Hamidin A, Azhar MZ, Noorjan KO, Salmiah MS, Bahariah K. Quality of life among patients with hematological cancer in a Malaysian hospital. Med J Malaysia. 2011 Jun;66(2):117-20. PMID 22106690
- [Result] Hansen DG, Larsen PV, Holm LV, Rottmann N, Bergholdt SH, Sondergaard J. Association between unmet needs and quality of life of cancer patients: a population-based study. Acta Oncol. 2013 Feb;52(2):391-9. doi: 10.3109/0284186X.2012.742204. Epub 2012 Dec 17. PMID 23244672
- [Result] Dietz JH Jr. Rehabilitation of the cancer patient. Med Clin North Am. 1969 May;53(3):607-24. No abstract available. PMID 4305950
- [Result] Banks E, Byles JE, Gibson RE, Rodgers B, Latz IK, Robinson IA, Williamson AB, Jorm LR. Is psychological distress in people living with cancer related to the fact of diagnosis, current treatment or level of disability? Findings from a large Australian study. Med J Aust. 2010 Sep 6;193(S5):S62-7. doi: 10.5694/j.1326-5377.2010.tb03931.x. PMID 21542449
- [Result] Kim YM, Kim DY, Chun MH, Jeon JY, Yun GJ, Lee MS. Cancer rehabilitation: experience, symptoms, and needs. J Korean Med Sci. 2011 May;26(5):619-24. doi: 10.3346/jkms.2011.26.5.619. Epub 2011 Apr 21. PMID 21532851
- [Result] Spill GR, Hlubocky FJ, Daugherty CK. Oncologists' and physiatrists' attitudes regarding rehabilitation for patients with advanced cancer. PM R. 2012 Feb;4(2):96-108. doi: 10.1016/j.pmrj.2011.08.539. PMID 22373458
- [Result] Handberg C, Jensen CM, Maribo T. Lack of Needs Assessment in Cancer Survivorship Care and Rehabilitation in Hospitals and Primary Care Settings. J Clin Med Res. 2017 Oct;9(10):864-871. doi: 10.14740/jocmr3160w. Epub 2017 Sep 1. PMID 28912923